CLINICAL TRIAL: NCT01128881
Title: IMMUNINE - Purified Factor IX Concentrate Virus-Inactivated: A Phase 4, Prospective, Open-label Multicenter Study to Prospectively Document the Exposure of IMMUNINE and to Monitor FIX Inhibitors in Previously Treated Patients With Severe (FIX Level < 1%) or Moderately Severe (FIX Level <= 2%) Hemophilia B Who Are Planned to Enter BAX 326 Study 250901 to Investigate a New Recombinant FIX Concentrate
Brief Title: IMMUNINE Pre-Treatment Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050901; 2009-016719-39 (EudraCT Number)
Record Dates: First submitted 2010-05-07; First posted 2010-05-24 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — prothrombin complex concentrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMMUNINE (Experimental)
  Interventions: Biological: Factor IX Concentrate (purified, virus-inactivated)

INTERVENTIONS:
Biological: Factor IX Concentrate (purified, virus-inactivated) — Intravenous injection/infusion; dose for prophylaxis: 20-40 IU/kg bodyweight, twice weekly (which may be adjusted to the subject´s bleeding pattern and lifestyle); dose for bleeding episodes and surgery: according to the Summary of Product Characteristics and the Product Information Leaflet of the respective country.
  Other Names: IMMUNINE

SUMMARY:
The primary objective of this study is to prospectively document the exposure to IMMUNINE and to monitor FIX inhibitors over a period of approximately 20 to 50 exposure days while receiving prophylactic treatment in up to 50 previously treated patients (PTPs) aged 12-64 years and approximately 20 pediatric PTPs up to 11 years of age with severe (FIX level < 1%) or moderately severe (FIX level <= 2%) hemophilia B who are planned to enter BAX326 study 250901, provided all eligibility criteria are met.

In addition, this study will evaluate the efficacy, safety, immunogenicity, thrombogenicity, and health-related quality of life (HR QoL) of these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is up to 64 years old at the time of screening
* Subject and/or legal representative has/have provided signed informed consent
* Subject has severe (FIX level < 1%) or moderately severe (FIX level <= 2%) hemophilia B (based on the one stage activated partial thromboplastin time (aPTT) assay), as tested at screening at the central laboratory
* Subject is previously treated with plasma-derived or recombinant FIX concentrate(s), cryoprecipitate or fresh frozen plasma (FFP) for approximately 100-150 exposure days (EDs) if >= 6 years old, or 20-50 EDs if < 6 years old, and is planned to enter BAX326 study 250901. The number of EDs are derived from the subject's treatment regimen and his/her bleeding pattern
* Subject is willing to receive prophylactic treatment for the duration of the study
* Subject is immunocompetent as evidenced by a CD4 count >= 200 cells/mm(3)
* Subject is human immunodeficiency (HIV) negative or is HIV+ with a viral load < 200 particles/μL ~ < 400,000 copies/mL
* Female subject of childbearing potential, presents with a negative serum pregnancy test, and agrees to employ adequate birth control measures for the duration of the study
* Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* The subject has a detectable factor IX inhibitor at screening, with a titer >= 0.6 Bethesda Units (BU) as determined by the Nijmegen modification of the Bethesda assay in the central laboratory
* The subject has a history of factor IX inhibitors with a titer >= 0.6 BU (as determined by the Nijmegen modification of the Bethesda assay or the assay employed in the respective local laboratory) at any time prior to screening
* The subject has a history of allergic reaction, eg, anaphylaxis, following exposure to factor IX concentrate(s)
* The subject has a known hypersensitivity to hamster proteins
* The subject has evidence of a thrombotic disease, fibrinolysis or disseminated intravascular coagulation (DIC)
* The subject is scheduled for elective surgery, unless the surgery is medically required within the anticipated study period
* The subject has an abnormal renal function (serum creatinine > 1.5 times the upper limit of normal)
* The subject has severe chronic liver disease as evidenced by, but not limited to, any of the following: International Normalized Ratio (INR) exceeding the upper limit of normal (ULN), hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices
* The subject has active hepatic disease with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels >= 5 times the upper limit of normal. During the study, subjects with chronic hepatitis B or C may have fluctuations of up to 5 times the upper limit of normal but will not require discontinuation.
* The subject has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia B
* The subject's platelet count is < 100,000/mL
* The subject has a clinically significant medical, psychiatric, or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect subject's safety or compliance
* The subject is currently receiving, or is scheduled to receive during the course of the study, an immunomodulating drug other than anti-retroviral chemotherapy (eg, α-interferon, corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 mg/day)
* The subject is unwilling to consider further participation in BAX 326 (rFIX) pivotal study 250901 or BAX 326 pediatric study
* The subject has participated in another investigational study within 30 days of enrollment or is scheduled to participate in another clinical study involving an investigational product (IP) or investigational device during the course of this study
* The subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study.

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2010-05-31 (Actual); Primary Completion 2012-08-28 (Actual); Study Completion 2012-08-28 (Actual)

PRIMARY OUTCOMES:
Hemostatic Efficacy | 28 months
  * Number of IMMUNINE infusions required to achieve adequate hemostasis for each bleeding episode
  * Overall hemostatic efficacy rating of IMMUNINE for all bleeding episodes (scale of excellent, good, fair, none)
  * Annualized bleeding rate
  * Consumption of IMMUNINE
  * Number of infusions per month and per year (prophylaxis and on-demand)
  * Weight-adjusted consumption of IMMUNINE per event (prophylaxis, on-demand), per month and per year

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (18):
- Argentina (2):
  - Hospital JR Vidal (Servicio de Hemotologie - Area de Investiagacion, Corrientes
  - Instituto de Hemofilia y Medicina Clinica Rubén Dávoli, Rosario
- Brazil (2):
  - Hospital do apoio de Brasilia, Distrito Federal
  - UNIFESP - Universidade Estadual de Sáo Paulo, Sáo Paulo
- Specialized Haematological Hospital "Joan Pavel", Sofia, Bulgaria
- Chile (2):
  - Hospital Dr. Sotero del Rio, Santiago
  - Hospital san José, Centro de Hemofilia, Santiago
- Centro Medico Imbanaco, Cali, Colombia
- Klinika detske hematologie a onkologie UK, Prague, Czechia
- Poland (4):
  - Hematology and Transplantology Clinic, University Clinic Centre - Medical University Hospital, Gdansk
  - Medical College of the Jagiellonian University, Krakow
  - Medical University Lodz, Department of Hematology, Lodz
  - Institute of Haematology and Transfusion, Warsaw
- Romania (2):
  - Prof. Dr. C. T. Nicolau National Institute for Transfusional Hematology, Bucharest
  - Louis Turcanu Emergency Clinical Children´s Hospital, Timișoara
- Russia (2):
  - Hematology Research Center RAMS, Department of Hemophilia and Other Coagulopathies, Moscow
  - Republican Center for Hemophilia Treatment, Outpatient Clinic No. 37, Saint Petersburg
- State Institution "Institute of Blood Pathology and Transfusion Medicine of Academy of Medical Sciences of Ukraine", Lviv, Ukraine